CLINICAL TRIAL: NCT02075697
Title: Spanish Registry of Systemic Treatments in Psoriasis
Acronym: Biobadaderm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Academia Española de Dermatología (Other)
Collaborators: Spanish Agency of Medicines and Health Products (Other Government); Janssen, LP (Industry); Merck Sharp & Dohme LLC (Industry); Pfizer (Industry); AbbVie (Industry); Eli Lilly and Company (Industry); Novartis (Industry); Boehringer Ingelheim (Industry); Bristol-Myers Squibb (Industry); UCB Pharma (Industry); Almirall, SAS (Industry); Amgen (Industry); LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: Biobadaderm; Biobadaderm (Registry Identifier: Biobadaderm)
Record Dates: First submitted 2013-01-03; First posted 2014-03-03 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Psoriasis
Keywords: psoriasis; biologic therapy; infliximab; etanercept; efalizumab; adalimumab; ustekinumab; methotrexate; cyclosporine; acitretin
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- New drugs: Cohort exposed to biologic therapy, apremilast or fumarates
- Classic systemic therapy: Non-biological systemic treatment (methotrexate, cyclosporine and acitretin) Phototherapy was accepted as systemic therapy only in the small group of patients retrospectively included(PUVA, UVB 311).

SUMMARY:
The purpose of Biobadaderm is a to study the safety of systemic therapy in psoriasis.

DETAILED DESCRIPTION:
The Spanish Registry for Adverse Events of Biological Therapies in Dermatology (BIOBADADERM) was launched in October 2008, as a pharmacovigilance effort for psoriatic patients. The registry is managed by the Foundation of the Spanish Academy of Dermatology and Venereology (AEDV). BIOBADADERM has been promoted by the AEDV, in collaboration with the Spanish Agency for Medicines and Health Products (AEMPS) and the Research Unit of the Spanish Foundation of Rheumatology (FER) and the Research Unit of the Fundacion AEDV. BIOBADADERM is part of PSONET, a European network for sharing data from records of patients treated with biologics.

BIOBADADERM is a prospective cohort of patients receiving biologic drugs that can be compared with another cohort of patients receiving other systemic treatments. One of the cohorts is made up of all consecutive psoriasis patients who begin any biological therapy (including infliximab (INF), etanercept (ET), efalizumab (EFA), adalimumab (ADA), rituximab (RTX) and ustekinumab (UTK)) in each centre. The control cohort consists of psoriasis patients who begin, for the first time, a nonbiologic systemic treatment (methotrexate, cyclosporine or acitretin).

The objectives of BIOBADADERM are:

* Identify adverse events (AEs) occurring during the relevant treatment with biologic therapies, and estimate their frequency;
* Identify unexpected AEs, particularly those that may occur after long periods of exposure;
* Identify relevant AEs that arise after discontinuation of treatment;
* Estimate the relative risk of developing AEs with biologic therapies in patients with psoriasis compared to psoriatic patients exposed to other systemic (non-biological); and
* Identify risk factors for AEs in patients with these treatments.

Data were initially collected retrospectively in hospitals with a list of all patients who had received biologic drugs between 1 January 2005 and 30 October 2008 and check-ups with a frequency of at least every 6 months. Since 2008, data have been captured prospectively.

The database includes demographic, diagnostic and comorbidity data, the treatments performed, the duration of these treatments and the adverse effects that arise (coded using MedDRA). In its first year, 632 patients from 12 centers participated with BIOBADADERM. In October 2012 the registry had data from 1,793 patients, which includes 946 patients on biologic treatments and 847 patients on non-biologic systemic treatments.

Data for each patient have been reversibly anonymized and entered into a database. Data are entered over the Internet (http://biobadaser.ser.es/biobadaderm/). The data are stored in the Research Department of the Spanish Rheumatology Foundation.

The included data are continually revised online by a study monitor to verify consistency, comprehensiveness, and absence of anomalies. A follow-up visit is made every year during which a sample of the the data in the database are compared with those in the clinical records.

Sample size was calculated to give, after 5 years, 80% power and using alfa level= 0.05, to detect a rate ratio of 2 in events with 4.1 cases per 1000 person-years, or a rate ratio of 5 in events with 0.5 cases per 1000 person-years. Further calculations are available in the study protocol (https://biobadaser.ser.es/biobadaderm/index.html).

Default value in each variable is "missing". Plans for missing data in analysis depend on the aim of analysis but with a preference for the most conservative ( in terms of patient safety) analysis.

Analysis consists of description of rates, rate ratios and adjusted rate ratios (adjusted for possible confounders, age always included).

ELIGIBILITY:
Inclusion Criteria:

* For biologics group: all consecutive psoriasis patients who begin any biological therapy
* For classic systemic group: the next psoriasis patients who begin, for the first time, a nonbiologic systemic treatment (after including a patient in the biologics group)

Exclusion Criteria:

* Intention of moving to a different geographic area in the next three months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Psoriasis patients requiring systemic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2008-10; Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | an expected mean follow-up of 5 years
  Rates and trate ratio compared to other drugs. Lag windows used to link events and therapy are described in the study web site.

SECONDARY OUTCOMES:
Other adverse events leading to changes in drug therapy or unexpected visits to health provider | an expected mean follow-up of 5 years
  Rate

OTHER OUTCOMES:
Mortality | an expected mean follow-up of 5 years
  Rate

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Daudén, PhD, Principal Investigator — Hospital de La Princesa- Madrid
Locations (13):
- Spain (13):
  - Hospital Universitari German Trias y Pujol., Badalona, Barcelona
  - Fundación Hospital Alcorcón, Alcorcón, Madrid
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clinic, Barcelona
  - Hospital del Mar. IMAS, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario de Gran Canaria Dr Negrín, Las Palmas
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena de Sevilla, Seville
  - Hospital General Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rivera R, Garcia-Doval I, Carretero G, Dauden E, Sanchez-Carazo J, Ferrandiz C, Herrera E, Alsina M, Ferran M, Lopez-Estebaranz JL, Gomez F, Herranz JM, Carrascosa JM, Vanaclocha F; miembros del grupo BIOBADADERM. [BIOBADADERM, the Spanish Registry of Adverse Events Associated with Biologic Drugs in Dermatology: first report]. Actas Dermosifiliogr. 2011 Mar;102(2):132-41. doi: 10.1016/j.ad.2010.10.016. Epub 2011 Mar 4. Spanish. PMID 21377137
- [Result] Garcia-Doval I, Carretero G, Vanaclocha F, Ferrandiz C, Dauden E, Sanchez-Carazo JL, Alsina M, Herrera-Ceballos E, Gomez-Garcia FJ, Ferran M, Lopez-Estebaranz JL, Hernanz JM, Belinchon-Romero I, Vilar-Alejo J, Rivera R, Carrascosa JM, Carazo C. Risk of serious adverse events associated with biologic and nonbiologic psoriasis systemic therapy: patients ineligible vs eligible for randomized controlled trials. Arch Dermatol. 2012 Apr;148(4):463-70. doi: 10.1001/archdermatol.2011.2768. PMID 22508869
- [Result] Sanchez-Moya AI, Garcia-Doval I, Carretero G, Sanchez-Carazo J, Ferrandiz C, Herrera Ceballos E, Alsina M, Ferran M, Lopez-Estebaranz JL, Gomez-Garcia F, De la Cueva Dobao P, Carrascosa JM, Vanaclocha F, Belinchon I, Peral F, Dauden E; BIOBADADERM Study Group. Latent tuberculosis infection and active tuberculosis in patients with psoriasis: a study on the incidence of tuberculosis and the prevalence of latent tuberculosis disease in patients with moderate-severe psoriasis in Spain. BIOBADADERM registry. J Eur Acad Dermatol Venereol. 2013 Nov;27(11):1366-74. doi: 10.1111/jdv.12011. Epub 2012 Nov 8. PMID 23134268
- [Result] Carrascosa JM, Vilavella M, Garcia-Doval I, Carretero G, Vanaclocha F, Dauden E, Gomez-Garcia FJ, Herrera-Ceballos E, De la Cueva Dobao P, Belinchon I, Sanchez-Carazo JL, Alsina M, Lopez-Estebaranz JL, Ferran M, Peral F, Torrado R, Rivera R, Jimenez-Puya R, Mendiola MV, Ferrandiz C; BIOBADADERM Study Group. Body mass index in patients with moderate-to-severe psoriasis in Spain and its impact as an independent risk factor for therapy withdrawal: results of the Biobadaderm Registry. J Eur Acad Dermatol Venereol. 2014 Jul;28(7):907-14. doi: 10.1111/jdv.12208. Epub 2013 Jul 15. PMID 23848131
- [Result] Garcia-Doval I, Rustenbach SJ, Stern R, Dam TN, Cohen AD, Baker C, Spuls PI, Naldi L; Psonet Network. Systemic psoriasis therapy shows high between-country variation: a sign of unwarranted variation? Cross-sectional analysis of baseline data from the PSONET registries. Br J Dermatol. 2013 Sep;169(3):710-4. doi: 10.1111/bjd.12344. No abstract available. PMID 23551034
- [Result] Medina C, Carretero G, Ferrandiz C, Dauden E, Vanaclocha F, Gomez-Garcia FJ, Herrera-Ceballos E, De la Cueva-Dobao P, Belinchon I, Sanchez-Carazo JL, Alsina M, Lopez-Estebaranz JL, Ferran M, Carrascosa JM, Torrado R, Argila D, Rivera R, Jimenez-Puya R, Garcia-Doval I; BIOBADADERM Study Group. Safety of classic and biologic systemic therapies for the treatment of psoriasis in elderly: an observational study from national BIOBADADERM registry. J Eur Acad Dermatol Venereol. 2015 May;29(5):858-64. doi: 10.1111/jdv.12688. Epub 2014 Sep 3. PMID 25185962
- [Result] Carretero G, Ferrandiz C, Dauden E, Vanaclocha Sebastian F, Gomez-Garcia FJ, Herrera-Ceballos E, De la Cueva-Dobao P, Belinchon I, Sanchez-Carazo JL, Alsina-Gibert M, Lopez-Estebaranz JL, Ferran M, Torrado R, Carrascosa JM, Carazo C, Rivera R, Jimenez-Puya R, Garcia-Doval I; BIOBADADERM Study Group. Risk of adverse events in psoriasis patients receiving classic systemic drugs and biologics in a 5-year observational study of clinical practice: 2008-2013 results of the Biobadaderm registry. J Eur Acad Dermatol Venereol. 2015 Jan;29(1):156-63. doi: 10.1111/jdv.12492. Epub 2014 Mar 31. PMID 24684267
- [Result] Garcia-Doval I, Perez-Zafrilla B, Ferrandiz C, Carretero G, Dauden E, de la Cueva P, Gomez-Garcia FJ, Herrera-Ceballos E, Belinchon-Romero I, Sanchez-Carazo JL, Lopez-Estebaranz JL, Alsina M, Ferran M, Torrado R, Carrascosa JM, Rivera R, Vanaclocha F; BIOBADADERM Study Group. Development of clinical prediction models for good or bad response to classic systemic drugs, anti-TNFs, and ustekinumab in psoriasis, based on the BIOBADADERM cohort. J Dermatolog Treat. 2016;27(3):203-9. doi: 10.3109/09546634.2015.1088130. Epub 2015 Sep 25. PMID 26367799
- [Result] Sanz-Bueno J, Vanaclocha F, Garcia-Doval I, Torrado R, Carretero G, Dauden E, Patricia Ruiz-Genao D, Alsina-Gibert MM, Perez-Zafrilla B, Perez-Rial G, Rivera R; members of the BIOBADADERM group. Risk of Reactivation of Hepatitis B Virus Infection in Psoriasis Patients Treated With Biologics: A Retrospective Analysis of 20 Cases From the BIOBADADERM Database. Actas Dermosifiliogr. 2015 Jul-Aug;106(6):477-82. doi: 10.1016/j.ad.2015.01.010. Epub 2015 Mar 13. English, Spanish. PMID 25776200
- [Result] Carrascosa JM, Garcia-Doval I, Perez-Zafrilla B, Carretero G, Vanaclocha F, Dauden E, De la Cueva-Dobao P, Belinchon I, Alsina M, Lopez-Estebaranz JL, Ferran M, Torrado R, Rivera R, Carazo C, Barboza L, Ferrandiz C; BIOBADADERM Study Group. Use of off-label doses is frequent in biologic therapy for moderate to severe psoriasis: A cross-sectional study in clinical practice. J Dermatolog Treat. 2015;26(6):502-6. doi: 10.3109/09546634.2015.1034070. Epub 2015 Apr 17. PMID 25886087
- [Result] Carrascosa JM, Rivera N, Garcia-Doval I, Carretero G, Vanaclocha F, Dauden E, Gomez-Garcia FJ, De-la-Cueva-Dobao P, Herrera-Ceballos E, Belinchon I, Alsina M, Sanchez-Carazo JL, Ferran M, Lopez-Estebaranz JL, Perez-Zafrilla B, Llamas M, Rivera R, Ferrandiz C; BIOBADADERM Study Group. Does the treatment ladder for systemic therapy in moderate to severe psoriasis only go up? The percentage of patients with severe psoriasis on biologics increases over time. Actas Dermosifiliogr. 2015 Oct;106(8):638-43. doi: 10.1016/j.ad.2015.04.013. Epub 2015 Jun 30. English, Spanish. PMID 26141003
- [Result] Ruiz-Genao D, Perez-Zafrilla B, Lopez-Estebaranz JL, Belinchon-Romero I, Carrascosa JM, Ferran M, Vanaclocha F, Herrera-Ceballos E, Garcia-Doval I; Biobadaderm Study Group. Possible paradoxical occurrence of inflammatory arthritis in patients with psoriasis treated with biologics: findings in the Biobadaderm cohort. Br J Dermatol. 2017 Mar;176(3):797-799. doi: 10.1111/bjd.14690. Epub 2016 Oct 17. No abstract available. PMID 27120993
- [Result] Garcia-Doval I, Hernandez MV, Vanaclocha F, Sellas A, de la Cueva P, Montero D; BIOBADADERM and BIOBADASER study groups. Should tumour necrosis factor antagonist safety information be applied from patients with rheumatoid arthritis to psoriasis? Rates of serious adverse events in the prospective rheumatoid arthritis BIOBADASER and psoriasis BIOBADADERM cohorts. Br J Dermatol. 2017 Mar;176(3):643-649. doi: 10.1111/bjd.14776. Epub 2016 Oct 3. PMID 27258623
- [Result] Davila-Seijo P, Dauden E, Carretero G, Ferrandiz C, Vanaclocha F, Gomez-Garcia FJ, Herrera-Ceballos E, De la Cueva-Dobao P, Belinchon I, Sanchez-Carazo JL, Alsina M, Lopez-Estebaranz JL, Ferran M, Torrado R, Carrascosa JM, Llamas M, Rivera R, Jimenez-Puya R, Garcia-Doval I; BIOBADADERM Study Group. Survival of classic and biological systemic drugs in psoriasis: results of the BIOBADADERM registry and critical analysis. J Eur Acad Dermatol Venereol. 2016 Nov;30(11):1942-1950. doi: 10.1111/jdv.13682. Epub 2016 Jun 22. PMID 27329511
- [Result] Davila-Seijo P, Dauden E, Descalzo MA, Carretero G, Carrascosa JM, Vanaclocha F, Gomez-Garcia FJ, De la Cueva-Dobao P, Herrera-Ceballos E, Belinchon I, Lopez-Estebaranz JL, Alsina M, Sanchez-Carazo JL, Ferran M, Torrado R, Ferrandiz C, Rivera R, Llamas M, Jimenez-Puya R, Garcia-Doval I; BIOBADADERM Study Group. Infections in Moderate to Severe Psoriasis Patients Treated with Biological Drugs Compared to Classic Systemic Drugs: Findings from the BIOBADADERM Registry. J Invest Dermatol. 2017 Feb;137(2):313-321. doi: 10.1016/j.jid.2016.08.034. Epub 2016 Sep 25. PMID 27677836
- [Result] Garcia-Doval I, Cohen AD, Cazzaniga S, Feldhamer I, Addis A, Carretero G, Ferrandiz C, Stern RS, Naldi L; Psonet Network. Risk of serious infections, cutaneous bacterial infections, and granulomatous infections in patients with psoriasis treated with anti-tumor necrosis factor agents versus classic therapies: Prospective meta-analysis of Psonet registries. J Am Acad Dermatol. 2017 Feb;76(2):299-308.e16. doi: 10.1016/j.jaad.2016.07.039. Epub 2016 Sep 29. PMID 27693008
- [Result] Davila-Seijo P, Garcia-Doval I, Naldi L, Cazzaniga S, Augustin M, Rustenbach SJ, Dauden E, Dam TN, Baker C, Spuls PI, Stern RS, Cohen AD. Factors Associated with Receiving Biologics or Classic Systemic Therapy for Moderate-to-Severe Psoriasis: Evidence from the PSONET Registries. Acta Derm Venereol. 2017 Apr 6;97(4):516-518. doi: 10.2340/00015555-2586. No abstract available. PMID 27882386
- [Result] Perez-Plaza A, Carretero G, Ferrandiz C, Vanaclocha F, Gomez-Garcia FJ, Herrera-Ceballos E, De la Cueva-Dobao P, Belinchon I, Sanchez-Carazo JL, Alsina M, Lopez-Estebaranz JL, Ferran M, Torrado R, Carrascosa JM, Llamas-Velasco M, Rivera R, Jimenez-Puya R, Garcia-Doval I, Descalzo MA; Biobadaderm Study Group. Comparison of phenotype, comorbidities, therapy and adverse events between psoriatic patients with and without psoriatic arthritis. Biobadaderm registry. J Eur Acad Dermatol Venereol. 2017 Jun;31(6):1021-1028. doi: 10.1111/jdv.14188. Epub 2017 Apr 12. PMID 28252811
- [Result] Belinchon I, Ramos JM, Carretero G, Ferrandiz C, Rivera R, Dauden E, De la Cueva-Dobao P, Gomez-Garcia FJ, Herrera-Ceballos E, Sanchez-Carazo JL, Lopez-Estebaranz JL, Alsina M, Ferran M, Torrado R, Carrascosa JM, Llamas-Velasco M, Ortiz PL, Garcia-Doval I, Descalzo MA; Biobadaderm Study Group. Adverse events associated with discontinuation of the biologics/classic systemic treatments for moderate-to-severe plaque psoriasis: data from the Spanish Biologics Registry, Biobadaderm. J Eur Acad Dermatol Venereol. 2017 Oct;31(10):1700-1708. doi: 10.1111/jdv.14314. Epub 2017 Jun 6. PMID 28485816
- [Result] Descalzo MA, Carretero G, Ferrandiz C, Rivera R, Dauden E, Gomez-Garcia FJ, de la Cueva P, Herrera-Ceballos E, Belinchon I, Lopez-Estebaranz JL, Alsina M, Sanchez-Carazo JL, Ferran M, Baniandres O, Carrascosa JM, Llamas-Velasco M, Ruiz-Genao D, Herrera-Acosta E, Munoz-Santos C, Garcia-Doval I; Biobadaderm Study Group. Change over time in the rates of adverse events in patients receiving systemic therapy for psoriasis: A cohort study. J Am Acad Dermatol. 2018 Apr;78(4):798-800. doi: 10.1016/j.jaad.2017.10.051. Epub 2017 Nov 13. No abstract available. PMID 29146129
- [Result] Garcia-Doval I, Descalzo MA, Mason KJ, Cohen AD, Ormerod AD, Gomez-Garcia FJ, Cazzaniga S, Feldhamer I, Ali H, Herrera-Acosta E, Griffiths CEM, Stern RS, Naldi L; Psonet Network. Cumulative exposure to biological therapy and risk of cancer in patients with psoriasis: a meta-analysis of Psonet studies from Israel, Italy, Spain, the U.K. and Republic of Ireland. Br J Dermatol. 2018 Oct;179(4):863-871. doi: 10.1111/bjd.16715. Epub 2018 Jul 24. PMID 29723914
- [Result] Carretero Hernandez G, Ferrandiz C, Rivera Diaz R, Dauden Tello E, de la Cueva-Dobao P, Gomez-Garcia FJ, Herrera-Ceballos E, Belinchon Romero I, Lopez-Estebaranz JL, Alsina Gibert M, Sanchez-Carazo JL, Ferran Farres M, Gonzalez Quesada A, Carrascosa Carrillo JM, Llamas-Velasco M, Mendiola Fernandez MV, Ruiz Genao D, Munoz Santos C, Garcia-Doval I, Descalzo MA; grupo de estudio de Biobadaderm. Description of Patients Treated with Biologic Drugs as First-Line Systemic Therapy in the BIOBADADERM Registry Between 2008 and 2016. Actas Dermosifiliogr (Engl Ed). 2018 Sep;109(7):617-623. doi: 10.1016/j.ad.2018.04.004. Epub 2018 Jun 7. English, Spanish. PMID 29887167
- [Result] Montes-Torres A, Aparicio G, Rivera R, Vilarrasa E, Marcellan M, Notario J, Soria C, Belinchon I, de la Cueva P, Ferran M, Carrascosa JM, Gomez FJ, Salgado L, Velasco M, Descalzo MA, Garcia-Doval I, Dauden E; ; the BIOBADADERM Study Group and Psoriasis Group of the AEDV. Safety and effectiveness of conventional systemic therapy and biological drugs in patients with moderate to severe psoriasis and HIV infection: a retrospective multicenter study. J Dermatolog Treat. 2019 Aug;30(5):461-465. doi: 10.1080/09546634.2018.1535690. Epub 2018 Nov 28. PMID 30307344
- [Result] Gonzalez-Cantero A, Carretero G, Rivera R, Ferrandiz C, Dauden E, de la Cueva P, Gomez-Garcia FJ, Belinchon I, Herrera-Ceballos E, Ruiz-Genao D, Ferran M, Alsina M, Sanchez-Carazo JL, Baniandres O, Sahuquillo-Torralba A, Rodriguez L, Vilar J, Garcia C, Carrascosa JM, Llamas-Velasco M, Herrera-Acosta E, Lopez-Estebaranz JL, Botella-Estrada R, Descalzo MA, Garcia-Doval I; BIOBADADERM Study Group. Women with moderate-to-severe psoriasis in Spain (BIOBADADERM registry) show more than a 50% reduction in age-adjusted fertility rate when compared with the general population. Br J Dermatol. 2019 Nov;181(5):1085-1087. doi: 10.1111/bjd.18164. Epub 2019 Aug 13. No abstract available. PMID 31127858
- [Result] Sahuquillo-Torralba A, Carretero G, Rivera R, Ferrandiz C, Dauden-Tello E, de la Cueva P, Gomez-Garcia FJ, Belinchon I, Herrera-Acosta E, Ruiz-Genao D, Ferran M, Alsina M, Sanchez-Carazo JL, Baniandres O, Fernandez-Freire LR, Vilar J, Garcia-Donoso C, Carrascosa JM, Llamas-Velasco M, Herrera-Ceballos E, Lopez-Estebaranz JL, Pujol-Marco C, Descalzo MA, Garcia-Doval I; Biobadaderm Study Group. The risk of urinary tract infections in patients with psoriasis on systemic medications in Biobadaderm Registry: A prospective cohort study. J Am Acad Dermatol. 2020 Mar;82(3):738-741. doi: 10.1016/j.jaad.2019.07.028. Epub 2019 Jul 13. No abstract available. PMID 31306726
- [Result] Echeverria-Garcia B, Nuno-Gonzalez A, Dauden E, Vanaclocha F, Torrado R, Belinchon I, Perez-Zafrilla B; Grupo de estudio BIOBADADERM. A Case Series of Patients With Psoriasis Exposed to Biologic Therapy During Pregnancy: The BIOBADADERM Register and a Review of the Literature. Actas Dermosifiliogr. 2017 Mar;108(2):168-170. doi: 10.1016/j.ad.2016.09.004. Epub 2016 Oct 17. No abstract available. English, Spanish. PMID 27765165
- [Result] Galiano Mejias S, Carretero G, Ferrandiz C, Vanaclocha F, Dauden E, Gomez-Garcia FJ, Herrera-Ceballos E, Belinchon-Romero I, Sanchez-Carazo JL, Lopez-Estebaranz JL, Alsina M, Ferran M, Torrado R, Carrascosa JM, Rivera R, Llamas-Velasco M, Jimenez-Puya R, Mendiola MV, Ruiz-Genao D, Descalzo MA, de la Cueva Dobao P; del grupo Biobadaderm. Management of Biologic Therapy in Moderate to Severe Psoriasis in Surgical Patients: Data From the Spanish Biobadaderm Registry. Actas Dermosifiliogr. 2017 Jan-Feb;108(1):52-58. doi: 10.1016/j.ad.2016.08.003. Epub 2016 Sep 20. English, Spanish. PMID 27658689
- See also: List of Biobadaderm publications — https://biobadaderm.fundacionpielsana.es/publicaciones.aspx